CLINICAL TRIAL: NCT03620994
Title: The Predictive Value of Alarm Symptoms in Patients With Irritable Bowel Syndrome Based on Rome IV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 20188517
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; alarm symptoms; Roman IV
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Irritable Bowel Syndrome: All patients who were satisfied with the inclusion criteria and exclusion criteria in the department of the second affiliated hospital of Xi'an JiaoTong University, Xijing Hospital ,Tangdu Hospital or affiliated hospital of Northwest University received investigation. Patients who participate in the study are determined on their own initiative, with full understanding and informedness.

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most commonly diagnosed functional bowel disorders (FBD). IBS is diagnosed by symptom-based criteria，while the available literature suggests that symptom-based diagnostic algorithms, which often used for clinical and research studies, have poor sensitivity. Although diagnostic algorithms can discriminate IBS from health or upper gastrointestinal tract conditions, studies do not provide convincing evidence that the criteria can discriminate IBS from organic disease of the colon. Rectal bleeding, anemia, weight loss, fever, family history of colon cancer, and age above 50 years are considered the warning signs of severe gastrointestinal disease. Colonoscopy is the most direct way to rule out organic colonic diseases. There is no consensus so far on whether patients with suspected IBS lacking warning signs need colonoscopy or not. In 2016, the Rome IV criteria was updated and published. However, there are few studies on the clinical practice based on Rome IV. The value of alarm symptoms in discriminating organic disease from functional disorders remains uncertain and further research is needed. To evaluate the predictive value of alarm symptoms of IBS patients based on Roman IV, the investigators designed this cross-sectional study.

DETAILED DESCRIPTION:
Functional bowel disorders (FBD) are a spectrum of chronic gastrointestinal (GI) disorders characterized by predominant symptoms or signs of abdominal pain bloating, distention, and/or bowel habit abnormalities, and the absence of obvious anatomic or physiologic abnormalities identiﬁed by routine diagnostic examinations, as deemed clinically appropriate. Irritable bowel syndrome (IBS) is one of the most commonly diagnosed functional bowel disorders (FBD). characterized by abdominal pain and bowel dysfunction, presenting as constipation, diarrhea, or alternating periods of both. Incidence rates of IBS are seldom calculated, and prevalence estimates fluctuate both between and within countries. A literature review by Sperber and colleagues suggests that a global prevalence rate could not be estimated owing to the heterogeneity of the studies. The pooled prevalence rate that the investigators cited for North America, Europe, Australia, and New Zealand was 8.1%. While IBS is not associated with increased mortality rates, it represents a significant burden on affected patients and society as a result of direct medical costs, lost productivity, and reduced health-related quality of life.

The development and persistence of IBS symptoms are understood to be multifactorial. Consequently, diagnosis and treatment are complicated clinical endeavors. IBS is diagnosed by symptom-based criteria, initially proposed by Manning and subsequently modified and quantified in the Rome I, II, and III criteria. However, the available literature suggests that symptom based diagnostic algorithms, although often used for clinical and research studies, have poor sensitivity. Although diagnostic algorithms can discriminate IBS from health or upper gastrointestinal tract conditions, studies do not provide convincing evidence that the criteria can discriminate IBS from organic disease of the colon. Therefore, in clinical practice, medical history should include evidence of organic disease (alarm symptoms) in addition to the main symptoms. Rectal bleeding, anemia, weight loss, fever, family history of colon cancer, and age above 50 years are considered the warning signs of severe gastrointestinal disease. Colonoscopy is the most direct way to rule out organic colonic diseases. It is an agreement that patients who meet Rome criteria on IBS with warning signs are strongly advised to perform colonoscopy to rule out severe colonic diseases such as inflammatory bowel disease (IBD) and colorectal cancer . The diagnostic sensitivity of symptom criteria on irritable bowel syndrome without colonoscopy is not more than 69.7% in patients with suspected irritable bowel syndrome lacking warning signs. There is no consensus so far on whether patients with suspected IBS lacking warning signs need colonoscopy or not. However, the value of alarm symptoms in discriminating organic disease from functional disorders remains uncertain and further research is needed, especially as alarm features are common.

In 2016, the Rome IV criteria was updated and published, in which IBS involved several changes. And there are currently few clinical studies based on Roman IV. This cross-sectional study was designed to evaluate the predictive value of alarm symptoms for IBS and organic bowel diseases and the difference in predictive value between different subtypes based on Roman IV.

Data collection：Basic information: name, gender, race, age, BMI index (height, weight), marital status ；Gastrointestinal symptoms: IBS-related symptoms，change in form of stool，duration and incidence of symptoms； Alarm Symptoms: Rectal bleeding (black stool, blood on toilet paper), anemia, weight loss, fever, nocturnal symptoms； Lifestyle habits: eating habits (spicy stimulation, dietary fiber), smoking, drinking, sleep quality, daily exercise time; Family history: colorectal cancer, inflammatory bowel disease, celiac disease, etc; Personal history: history of gastrointestinal infections, life emergency events; Test results: laboratory test results，colonoscopy results. The investigators obtained relevant information through consultation, telephone follow-up, questionnaire follow-up.Through endoscopy results to determine organic or functional diseases, benign or malignant, through contacts with the basic data, to determine the alarm symptoms. Further more, this study was proved by the ethical committee of second hospital of Xi'an jiaotong university.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of Irritable bowel syndrome symptoms，that is，recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria:

   Related to defecation;

   Associated with a change in frequency of stool;

   Associated with a change in form (appearance) of stool.

   （Criteria fulﬁlled for the last 3 months with symptom onset at least 6 months before diagnosis.）
2. Aged 18 years and older;
3. August 2018 to March 2019, patients went to the Gastroenterology clinics of the second affiliated hospital of Xi'an JiaoTong University, Xijing Hospital ,Tangdu Hospital or affiliated hospital of Northwest University , and received Colonoscopy;
4. Blood routine examination, fecal routine examination, and fecal occult blood test were conducted within 6 months.

Exclusion Criteria:

1. Previously diagnosed with diseases that better explain the participant's IBS symptoms (e.g. celiac disease, colorectal cancer, inflammatory bowel disease, microscopic colitis, lactose intolerance, bile acid malabsorption, intestinal tuberculosis, diverticulosis, ischemic enteritis, etc.);
2. Metabolic disease: uncontrolled thyroid disease and diabetes;
3. Severe neurological and psychiatric disorders, which may impede conduct of the clinical trial. These disorders include but are not limited to major depression with a high risk of suicidal behavior (i.e. intent or plan), alcohol or substance abuse/dependence, a lifetime history of psychosis;
4. Participant has an unstable severe extraintestinal medical condition (such as heart, liver, kidney and respiratory failure) with immediate or foreseeable treatment needs;
5. Previous major abdominal surgery that would have resulted in significant changes in the anatomy or physiology of the gastrointestinal tract, which can fully explain GI symptoms. Note: appendectomy, cholecystectomy, endoscopic polypectomy, endoscopic mucosal resection and endoscopic submucosal resection are not excluded criteria;
6. Were pregnant, might become pregnant, or were lactating;
7. Colonoscopy for structural evaluation of the GI tract in the past 6 months due to their IBS symptoms;
8. Taking anti-anxiety, anti-depressant drugs or intestinal sensitive antibiotics recently;
9. A current infection or infection of any type within the 2 weeks prior to evaluation that would obscure the presentation of IBS symptoms, in which case the assessment can be delayed until 2 weeks after full recovery;
10. Currently diagnosed malignancy, with exception of localized basal or squamous cell carcinomas of the skin which is completely removed. The so-called "current" means that the diagnosis of any malignancy (except basal cells or squamous cell carcinoma) that is active occurs within the first 12 months of enrollment;
11. Refusal to participate in this study or who cannot follow the research requirements for various reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From August 2018 to March 2019, patients went to the Gastroenterology clinics of the second affiliated hospital of Xi'an JiaoTong University, Xijing Hospital ,Tangdu Hospital or affiliated hospital of Northwest University who met the inclusion criteria were followed up.Subjects are voluntarily involved in the study, provided that they are fully understood and informed. The patients included in this study are all patients who underwent colonoscopy and signed an informed consent form for colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of organic bowel diseases | 6 months
  To collect the results of colonoscopy in patients who meet inclusion criteria, and to calculate the incidence of organic bowel diseases to analyze the predictive value of alarm symptoms.

SECONDARY OUTCOMES:
The incidence of organic bowel diseases in different subtypes of IBS | 6 months
  To collect the results of colonoscopy in patients who meet subtypes criteria, and to calculate the incidence of organic bowel diseases to compare the difference in predictive value of alarm symptoms for different subtypes of IBS.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Wang, MD, Study Director — The Second Affiliated Hospital of Xi'an Jiaotong University,Xi'an, Shanxi, China
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi’an, Shanxi, China